CLINICAL TRIAL: NCT06273124
Title: Open, Single Arm, Prospective, Multicenter Study of an Investigational Extended Wear Insulin Infusion Set During Home Use in People With Type 1 Diabetes
Brief Title: Investigational Extended Wear Insulin Infusion Set in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150-1261-00
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Type1diabetes

STUDY DESIGN:
Intervention Model Description: Device Extended Wear Infusion Set Each participant will wear each extended wear infusion set for up to 168 hours for 12 sequential wear periods.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- SteadiSet Extended Wear Infusion Set (Experimental): Each participant will be asked to wear the Investigational Extended Wear Infusion Set for up to 168 hours for 12 consecutive wear periods with the Tandem t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 or G7 sensor.
  Interventions: Device: SteadiSet Extended Wear Infusion Set

INTERVENTIONS:
Device: SteadiSet Extended Wear Infusion Set — Each participant will be given 12 Extended Wear Infusion Sets to wear over 12 wear periods up to 168 hours each.

SUMMARY:
The purpose of this study is to collect clinical data to support a 7-day wear of the Extended Wear Infusion Set (EWIS).

Participants will be asked to:

1. Wear the EWIS for up to 7 consecutive days for 12 consecutive wear periods
2. Perform blood glucose and ketone measurements if continuous glucose meter is ≥250mg/dL for one hour

DETAILED DESCRIPTION:
This is a multi-center, single-arm, prospective study of an extended wear infusion set in adults with Type 1 diabetes using a Tandem t:slim X2 insulin pump with Control-IQ technology with continuous Glucose Monitoring (CGM). Up to 300 participants across the United States age 18-80 will be enrolled in up to 20 investigational centers. Participants will change insulin cartridge every 48 to 72 hours as recommended by their health care provider. Participants will be expected to participate in the study for approximately 12-16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Age 18 to 80 years old inclusive
  2. Generally in good health, as determined by the investigator
  3. Living in the United States with no plans to move outside the United States during the study
  4. Diagnosis of T1D for at least 12 months
  5. Minimum of 6 months of insulin pump experience and at least 3 months of current experience with a Tandem pump
  6. Using Tandem t:slim X2 insulin pump with Control-IQ technology for a minimum of 1 month at the time of enrollment
  7. Minimum of 14 days of Control-IQ data immediately preceding screening that demonstrate pump use compliance, including at least 85% of time with Control-IQ technology active
  8. HbA1c <9.0% in the last 6 months.
  9. Willing to implement and adhere to pump alert/alarm settings on a study-provided pump as instructed during the study
  10. Willing to wear each investigational infusion set for up to 7 days during each of the 12 consecutive wear periods in the study
  11. Willing to perform blood ketone and blood glucose (fingerstick) measurements as directed using provided ketone and blood glucose meters and strips
  12. Access to internet for required periodic uploads of study device data
  13. BMI in the range 18-35 kg/m2, both inclusive
  14. Currently using one of the following insulins with no expectation of a need to change insulin type during the study:

      1. Humalog™* (insulin lispro)
      2. NovoLog™* (insulin aspart)
  15. Using Humalog™ insulin lispro or NovoLog™ insulin aspart for a minimum of 1 month at the time of enrollment
  16. Willing to change insulin cartridge every 48-72 hours, as recommended by patient's healthcare provider during the study
  17. Has routine access to a smart phone e.g., ability to receive text messages
  18. Has the ability to understand and comply with protocol procedures and to provide informed consent (i.e., English proficient in both verbal and written communication)

Exclusion Criteria:

1. Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
2. Female subject is pregnant, planning to become pregnant, or not using adequate method of contraception
3. Episodes of severe hypoglycemia in the last 6 months resulting in:

   1. Medical Assistance (i.e., paramedics, hospital evaluation or hospitalization)
   2. Loss of consciousness
   3. Seizures
4. One or more episodes of diabetic ketoacidosis (DKA) in the last 6 months requiring hospitalization
5. Currently on a ketogenic or low-carbohydrate diet of less than 60 grams of carbohydrates per day, or intending to begin one during the study period
6. Known cardiovascular disease considered to be clinically relevant by the investigator
7. Known history of any of the following conditions:

   1. Cushing's Disease
   2. Pancreatic islet cell tumor
   3. Insulinoma
   4. Lipodystrophy
   5. Extensive lipohypertrophy, as assessed by the investigator
8. Currently undergoing treatment with:

   1. Systemic oral or intravenous corticosteroids (current or within the last 8 weeks from screening),
   2. Thyroid hormones, unless use has been stable during the past 3 months
9. Significant history of any of the following, that in the opinion of the investigator would compromise safety or successful study participation:

   1. Alcoholism
   2. Drug abuse
10. Significant acute or chronic illness, that in the opinion of the investigator might interfere with safety or integrity of study results
11. Current participation in another clinical drug or device study
12. Immediate family member (spouse, biological or legal guardian, child, sibling, parent) who is a study site personnel directly affiliated with this study or who is an employee of Capillary Biomedical

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alayne Lehman, RN, MS, Study Director — Capillary Biomedical
Locations (15):
- United States (15):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Stanford University, Stanford, California
  - Barbara Davis Center, Aurora, Colorado
  - Endocrine Research Solutions, Roswell, Georgia
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Northwestern University, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - International Diabetes Center - HealthPartners Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mt. Sinai, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Texas Diabetes and Endocrinology, Austin, Texas
  - Rainier Clinical Research Center, Renton, Washington
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lal RA, Lum JW, Reed ZW, Kruger D, Reed JC 3rd, Weinstock RS, Carlson AL, Kudva YC, Liljenquist D, Cobry EC, Levister CM, Aleppo G, Chen J, Ahn DT, Hirsch IB, Putman MS, Broyles F, Pinsker JE, Romey M, Lehman A, Muchmore DB, Kollman C, Beck RW; CB1 Study Group. A Multicenter Study of an Investigational Extended Wear Insulin Infusion Set in Adults with Type 1 Diabetes. Diabetes Technol Ther. 2025 Aug 8. doi: 10.1177/15209156251364548. Online ahead of print. PMID 40780817

RESULTS

PARTICIPANT FLOW:
Groups:
- SteadiSet Extended Wear Infusion Set - Humalog: Each participant will be asked to wear the Investigational Extended Wear Infusion Set for up to 168 hours for 12 consecutive wear periods with the Tandem t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 or G7 sensor.
  Approximately half of the participants in the study were using Humalog insulin.
- SteaduSet Extended Wear Infusion Set - Novolog: Each participant will be asked to wear the Investigational Extended Wear Infusion Set for up to 168 hours for 12 consecutive wear periods with the Tandem t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 or G7 sensor.
  Approximately half of the participants in the study were using Novolog insulin.
Period: Overall Study
Arm/Group | SteadiSet Extended Wear Infusion Set - Humalog | SteaduSet Extended Wear Infusion Set - Novolog
Started | 128 | 132
Completed | 124 | 126
Not Completed | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SteadiSet Extended Wear Infusion Set - Humalog | SteaduSet Extended Wear Infusion Set - Novolog | Total
Number analyzed (Participants) | 128 | 132 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (16.0) | 46.8 (18.0) | 43.9 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 67 | 150
  Male | 45 | 65 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 124 | 125 | 249
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 115 | 125 | 240
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 128 | 132 | 260

OUTCOME MEASURES:

1. Primary Outcome: 7 Day Survival of Infusion Set for Primary Outcome Measure - Humalog
Description: 7-day infusion set survival for primary outcome reasons as defined in the protocol (Hyperglycemia and failure to respond to boluses, Hyperglycemia with ketones >1.0 mmol/L, or Investigator advised), for participants using Humalog.
Time Frame: 12 weeks
Population: To be considered for analysis in the primary outcome, participants had to have successfully inserted at least 6 sets per the study protocol.
Measure: Mean (Standard Error); unit: percentage of infusion set wears
Units Other Than Participants: Number of Infusion Sets
Arm/Group | SteadiSet Extended Wear Infusion Set - Humalog
Number analyzed (Participants) | 124
Number analyzed (Number of Infusion Sets) | 1500
percentage of infusion set wears | 95 (0.7)
Statistical Analysis 1: Comparison: SteadiSet Extended Wear Infusion Set - Humalog; Ninety-five percent confidence intervals for the 7-day survival rates and p-values for the survival probabilities being greater than 75% were calculated with a bootstrap to account for the correlated data from having each participant wear multiple infusion sets; Test type: Superiority; p < 0.001, Bootstrapping Kaplan-Meier estimates; Kaplan-Meier 7 Day Survival Estimate = 95, 95% CI 2-sided [94 to 97]

2. Primary Outcome: 7 Day Survival of Infusion Set for Primary Outcome Measure - Novolog
Description: 7-day infusion set survival for primary outcome reasons as defined in the protocol (Hyperglycemia and failure to respond to boluses, Hyperglycemia with ketones >1.0 mmol/L, or Investigator advised), for participants using Novolog.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of infusion set wears
Units Other Than Participants: Number of Infusion Sets
Groups:
- SteadiSet Extended Wear Infusion Set - Novolog: Each participant will be asked to wear the Investigational Extended Wear Infusion Set for up to 168 hours for 12 consecutive wear periods with the Tandem t:slim X2 insulin pump with Control-IQ technology, and wearing the Dexcom G6 or G7 sensor.
  Approximately half of the participants in the study were using Novolog insulin.
Arm/Group | SteadiSet Extended Wear Infusion Set - Novolog
Number analyzed (Participants) | 126
Number analyzed (Number of Infusion Sets) | 1527
percentage of infusion set wears | 95 (0.8)
Statistical Analysis 1: Comparison: SteadiSet Extended Wear Infusion Set - Novolog; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Bootstrapping Kaplan-Meier estimates; Kaplan-Meier 7 Day Survival Estimate = 95, 95% CI 2-sided [93 to 96]

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | SteadiSet Extended Wear Infusion Set - Humalog | SteaduSet Extended Wear Infusion Set - Novolog
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/128 | 1/132
Other Adverse Events (participants affected / at risk) | 14/128 | 29/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SteadiSet Extended Wear Infusion Set - Humalog (N=128) | SteaduSet Extended Wear Infusion Set - Novolog (N=132)
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Diabetic Ketoacidosis (Endocrine disorders) | 0 (0) | 0 (0)
Other Serious Adverse Event (General disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SteadiSet Extended Wear Infusion Set - Humalog (N=128) | SteaduSet Extended Wear Infusion Set - Novolog (N=132)
Abscess NOS (Infections and infestations) | 0 (0) | 1 (1)
Atopic dermatitis (Infections and infestations) | 0 (0) | 1 (2)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 4 (4)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cycling accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Erythematous conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hyperglycemia with or without Ketosis (Endocrine disorders) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 4 (4) | 1 (1)
Injection site discomfort (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0)
Injection site irritation (Infections and infestations) | 0 (0) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Localized superficial swelling, mass, or lump (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Medical device site inflammation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Neurologic disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Pain in face (General disorders) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5)
Skin abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 4 (4)
Sulfonamide allergy (Immune system disorders) | 0 (0) | 1 (1)
Vulval itching (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Yeast infection (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT06273124/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT06273124/SAP_001.pdf